CLINICAL TRIAL: NCT05908578
Title: Exercise Frequency During Endurance Training: Cardiorespiratory, Hematological, and Muscle Oxidative Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Tom Tripp, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REB23-0467
Record Dates: First submitted 2023-05-28; First posted 2023-06-18 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Exercise Training
Keywords: Exercise; Muscle, Striated; Blood; Erythrocytes; Cardiorespiratory Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will undergo the same baseline testing before being pseudo-randomly (block randomization) allocated to one of two groups, each following a different exercise training program for eight weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Frequency Training (Active Comparator): Exercise performed on a stationary bike four times per week. Total weekly exercise volume (the product of intensity, duration, and frequency) will be matched between groups. Intensity will be the same, so the high-frequency group will perform half the duration of exercise in each session compared to the low-frequency group.
  Interventions: Other: High Frequency Exercise Training
- Low-Frequency Training (Experimental): Exercise performed on a stationary bike two times per week. Total weekly exercise volume (the product of intensity, duration, and frequency) will be matched between groups. Intensity will be the same, so the low-frequency group will perform double the duration of exercise in each session compared to the high-frequency group.
  Interventions: Other: Low Frequency Exercise Training

INTERVENTIONS:
Other: High Frequency Exercise Training — Two sessions per week of high-intensity interval training (30 min each) and two sessions per week of continuous endurance exercise (30 min each). All exercise sessions will be performed on a stationary bike under supervision by an investigator.
  Arms: High-Frequency Training
Other: Low Frequency Exercise Training — One session per week of high-intensity interval training (60 min) and one session per week of continuous endurance exercise (60 min). All exercise sessions will be performed on a stationary bike under supervision by an investigator.
  Arms: Low-Frequency Training

SUMMARY:
The goal of this interventional study is to compare training for different numbers of days each week in healthy, young individuals. The main questions it aims to answer are:

* Does exercising less often improve endurance fitness as much as exercising more often?
* Are endurance fitness improvements caused by improvements in the muscle and blood?

Participants will train on a stationary bike for eight weeks. Researchers will measure the participants endurance fitness, as well as muscle and blood characteristics, before and after training to look for improvements from the training protocols.

Researchers will compare low-frequency exercise (two times per week) and high-frequency exercise (four times per week) to see if they each improve endurance fitness.

DETAILED DESCRIPTION:
Questions and Hypotheses:

The primary research question of this study is "Does exercising less frequently lead to improvements in aerobic fitness that are not worse than the improvements from exercising more frequently, when total exercise volume and exercise intensity are matched?" The secondary research questions of this study are: "Does exercising less frequently lead to similar improvements in hemoglobin mass, neuromuscular fatigue resistance, and skeletal muscle oxidative capacity compared to exercising more frequently, when total exercise volume and exercise intensity are matched?" The investigators hypothesize that the "weekend warrior" training program will induce improvements in cardiorespiratory fitness that are not worse than the improvements elicited by the standard training protocol. The investigators hypothesize that these improvements will be driven by similar improvements in markers of skeletal muscle mitochondrial content, and hemoglobin mass, and neuromuscular fatigue resistance between both training protocols.

Study Design and Methods:

32 participants total (16 female, 16 male; 8 per sex per group) will be randomized to either the low- or high-frequency training groups and will undergo physiological testing at baseline, after 4 weeks, and after 8 weeks of training. The sample size of 32 was calculated based on an alpha of 0.05, a power of 0.90, a group allocation ratio of 1:1, and a dropout rate of 20%. As this study is using non-inferiority testing, the investigators also set the allowable difference to 0 (the null hypothesis), the standard deviation for change in the primary outcome to 3 (based on data from a recently completed study), and the non-inferiority margin to 3.5 mL/kg/min, which is equivalent to 1 metabolic equivalent of task unit (MET), a standard unit for assessing cardiorespiratory fitness that is often considered to have clinical significance.

The low- and high-frequency groups will perform exercise two or four days per week, respectively. The intensity and duration of training sessions will increase throughout the study to ensure the training stimulus is maintained as participants become fitter. Training intensities will be individualized based on exercise testing.

The investigators will measure (i) maximal oxygen uptake (V̇O2max) and ventilatory thresholds with an incremental exercise test; (ii) substrate oxidation and neuromuscular fatigue development during 30 minutes of constant work rate cycling in the heavy intensity domain, (iii) time to task failure at 80% of peak power output (i.e., "performance") following this prolonged exercise bout; (iv) hemoglobin mass with the carbon monoxide rebreathing technique; (v) non-invasive skeletal muscle oxidative capacity using near-infrared spectroscopy (NIRS). Throughout training, perceptual responses including rating of perceived exertion and rating of general fatigue will be recorded, as well as exercising heart rate and heart rate variability.

In total, participants in the high-frequency group will visit the laboratory 25 times and participants in the low-frequency group will visit the laboratory 40 times. For both groups, the total time commitment is ~37 hours spread over 12 weeks.

Training Programs:

Participants in the high-frequency and low-frequency training groups will visit the laboratory 31 and 16 times, respectively, to complete their exercise training. In total, with conservative rounding to the nearest half hour, participants will train for ~23 hours over 8 weeks.

Participants in the low-frequency group will complete 2 training sessions per week, whereas participants in the high-frequency group will complete 4 training sessions per week. To ensure that training volume is equal across groups, the low-frequency group will perform the same training sessions as the high-frequency group; however, they will perform them "back-to-back" each day. All exercise training will be based on the results of individual exercise tests.

For high-intensity interval training (HIIT), participants will perform 4 min of severe intensity exercise followed by 3 min of moderate intensity exercise. Each HIIT workout will be preceded by an 8-min warm-up. For the low-frequency group, the two HIIT workouts will be performed on the same day, but they will be interspersed by the same 8-min warm-up to ensure the total volume of exercise is equal between groups.

For the continuous training (CONT), participants will cycle at an intensity equal to ~50% of the difference between the gas exchange threshold and the respiratory compensation point. All CONT workouts will be preceded by the same 8-min warm-up. For the low-frequency group, the two CONT workouts will be performed on the same day, but they will be interspersed by the same 8-min warm-up to ensure the total volume of exercise is equal between groups.

Training load will remain constant for two weeks before either increasing in duration (week 3 and week 7) or intensity (week 5). The increase in intensity will be based on the mid-point V̇O2max test, which takes the place of 1 unit of CONT training for both groups.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent
* complete and pass the Get Active Questionnaire (GAQ), a physical activity readiness screening tool

Exclusion Criteria:

* classified as obese (BMI > 30 kg/m^2)
* taking medications that are known to affect cardiovascular and/or metabolic responses to exercise (including but not limited to beta-blockers, anti-inflammatories, anti-coagulants, insulin, etc.)
* dieting for weight loss or following a low carbohydrate diet
* smoking or using tobacco products within the previous year
* consuming excessive amounts of alcohol (>21 units/week)
* having known health problems such as renal or gastrointestinal disorders, metabolic disease, heart disease, vascular disease, arthritis, diabetes, respiratory disease, uncontrolled blood pressure, dizziness, thyroid problems, or any other health conditions that may confound results
* having orthopedic issues that limit exercise performance
* using an investigational drug product within the last 30 days
* are pregnant
* have donated blood in the previous 90 days
* being highly trained or engaging in training more than 4 times per week
* do not understand English

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline maximal oxygen uptake (VO2max) after 8 weeks of training | 8 weeks
  Change in maximal oxygen uptake determined using an incremental exercise test on a cycle ergometer, measured after 8 weeks of training relative to baseline

SECONDARY OUTCOMES:
Change from baseline near-infrared spectroscopy (NIRS)-derived oxidative capacity of the vastus lateralis muscle after 8 weeks of training | 8 weeks
  Non-invasive measure of muscle ability to use oxidative phosphorylation, measured using near-infrared spectroscopy on the surface of the skin. Measure is the change from baseline after 8 weeks of training.
Change from baseline hemoglobin mass after 8 weeks of training | 8 weeks
  Total hemoglobin mass determined through dilution of carbon monoxide in the blood. Measure is the change from baseline after 8 weeks of training
Change from baseline gas exchange threshold after 8 weeks of training | 8 weeks
  Ventilatory threshold during exercise that demarcates the moderate and heavy intensity domains. Expressed in absolute terms (L/min of O2) and relative to body mass (mL/min/kg) and lean body mass (mL/min/kg). Measure is the change from baseline after 8 weeks of training.
Change from baseline respiratory compensation point after 8 weeks of training | 8 weeks
  Ventilatory threshold during exercise that demarcates the heavy and severe intensity domains. Expressed in absolute terms (L/min of O2) and relative to body mass (mL/min/kg) and lean body mass (mL/min/kg). Measure is the change from baseline after 8 weeks of training.
Change from baseline peak power output after 8 weeks of training | 8 weeks
  Maximum power output achieved during the incremental cycling test. Measure is the change from baseline after 8 weeks of training
Change in time to task failure after 8 weeks of training | 8 weeks
  Cycling time completed at 85% of peak power output during the performance test. Measure is the change from baseline after 8 weeks of training.
Change in quadriceps maximal voluntary contraction (MVC) force decline in response to the same absolute exercise task, after 8 weeks of training | 8 weeks
  Exercise induces a decrease in maximal voluntary contraction (MVC) force of the quadriceps muscle group. The decline in MVC force in response to the same absolute exercise task (i.e., the same duration and power output) will be compared to baseline after 8 weeks of training.
Change in quadriceps maximal voluntary contraction (MVC) force decline in response to the same relative exercise task, after 8 weeks of training | 8 weeks
  Exercise induces a decrease in maximal voluntary contraction (MVC) force of the quadriceps muscle group. The decline in MVC force in response to the same relative exercise task (i.e., the same duration and percentage of lactate threshold) will be compared to baseline after 8 weeks of training.

CONTACTS AND LOCATIONS:
Overall Officials: Martin J MacInnis, PhD, Principal Investigator — University of Calgary
Locations (1):
- Human Performance Lab, University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tripp TR, Ghitter RS, Kontro H, Hargrave SJ, Gibala MJ, Aboodarda SJ, MacInnis MJ. Cardiorespiratory Fitness Improvements Following Low-Frequency Training Are Not Inferior to High-Frequency Training Matched for Intensity and Volume. Scand J Med Sci Sports. 2025 Feb;35(2):e70024. doi: 10.1111/sms.70024. PMID 39921357